CLINICAL TRIAL: NCT04263129
Title: Tracheobronchial Bioengineering Using Aortic Matrices
Brief Title: Tracheobronchial Bioengineering Using Aortic Matrices for Airway Reconstruction
Acronym: TRITON
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: TRITON
Record Dates: First submitted 2019-11-22; First posted 2020-02-10 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Tracheal Disease
Keywords: artificial trachea; tracheal reconstruction; bronchial reconstruction
MeSH Terms: conditions — Tracheal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Tracheal, carinal or bronchial transplantation using a stented cryopreserved aortic — Radical resection of the lesions was performed using standard surgical techniques. After resection, airway reconstruction was performed using a human cryopreserved (-80°C) aortic allograft, which was not matched by the ABO and leukocyte antigen systems. To prevent airway collapse, a custom-made stent was inserted into the allograft. In patients with proximal lung tumors, the lung-sparing intervention of bronchial transplantation was used.

SUMMARY:
A technic of tracheal, carinal or bronchial transplantation using a stented cryopreserved aortic has been implemented by Pr E. Martinod in his thoracic surgery dept. The purpose of this study is to analyze the records of all the patients who have benefited from this treatment.

DETAILED DESCRIPTION:
In the context of end-stage tracheobronchial disease (in particular tracheal or carinal indication) this technic propose a therapeutic alternative, in the context of bronchial replacement it allows to avoid pneumonectomy.

The advantages are to reduce mortality at 90 days, functional consequences and long-term complications.

In this observationnel study, data were collected prospectively in the medical records of all patients who have undergone a trachea or artificial bronchus transplant.

ELIGIBILITY:
Inclusion Criteria:Eligible patients were treated by human cryopreserved (-80°C) aortic allograft after undergoing a standard preoperative evaluation and cardiopulmonary tests. A multidisciplinary team approve d the treatment based on the following criteria: Patients (1) had proximal lung tumors requiring a surgical resection (pneumonectomy, carinal resection, or sleeve lobectomy) that may or may not have been treated with neoadjuvant chemotherapy and had adequate or compromised preoperative lung function tests; or (2) had significant major malignant or benign lesions of the trachea and bronchi untreated with conventional therapeutic approaches, and (3) have signed an informed consent form for this specific surgical intervention.

Exclusion Criteria:Patients were not treated by human cryopreserved (-80°C) aortic allograft if they :

(1) had a lung tumor requiring a standard lobectomy; (2) had nonresectable major locally invasive tumors; (3) had contralateral lymph node invasion; (4) had metastatic disease with the exception of a unique resectable brain metastasis; (5) had tracheal lesions requiring standard resection with direct anastomosis; (6) had an iodine allergy; or (7) received a preoperative evaluation indicating an inability to undergo a standard lobectomy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients treated by human cryopreserved (-80°C) aortic allograft in thoracic surgery dept of Avicenne Hospital, Bobigny, France
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Assessment of survival at 3 months | 3 months
  Rate of death at 3 months

SECONDARY OUTCOMES:
Assessment of survival at 12 months | 12 months
  Rate of death at 12 months
Assessment of survival at 60 months | 60 months
  Rate of death at 60 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital AVICENNES Service de Chirurgie Thoracique, Bobigny, France

REFERENCES:
- [Derived] Martinod E, Onorati I, Radu DM, Santos Portela AM, Peretti M, Bardet J, Maiolino E, Lo Torto S, Uzunhan Y, Freynet O, Chouahnia K, Duchemann B, Brillet PY, Clero D, Juvin C, Lebreton G, Rouard H, Kabbani J, Maurer C, Gauthier A, Mangiapan G, Dutau H, Marquette CH, Malet J, Deslee G, Galvaing G, Chadeyras JB, Tronc F, Gandher C, Buffet C, Bensidhoum M, Miyara M, Dard N, Besnard V, Planes C, Tresallet C, Fournier C, Venissac N, Huet O, Beloucif S, Vicaut E. Tracheobronchial Replacement Using Cryopreserved Aortic Allografts: Results in 50 Patients (TRITON-01 Registry). Eur J Cardiothorac Surg. 2026 Jan 6;68(1):ezaf445. doi: 10.1093/ejcts/ezaf445. PMID 41390914
- [Derived] Onorati I, Radu DM, Portela AMS, Peretti M, Guiraudet P, Bardet J, Freynet O, Didier M, Uzunhan Y, Chouahnia K, Duchemann B, Bourinet V, Dutau H, Berthet JP, Marquette CH, Tronc F, Sanchez ML, Tresallet C, Fournier C, Venissac N, Miyara M, Vicaut E, Martinod E. Preliminary results in tracheal replacement using stented aortic matrices for primary extensive tracheal cancer. JTCVS Tech. 2023 Jun 23;21:227-236. doi: 10.1016/j.xjtc.2023.05.021. eCollection 2023 Oct. PMID 37854807
- [Derived] Martinod E, Radu DM, Onorati I, Portela AMS, Peretti M, Guiraudet P, Destable MD, Uzunhan Y, Freynet O, Chouahnia K, Duchemann B, Kabbani J, Maurer C, Brillet PY, Fath L, Brenet E, Debry C, Buffet C, Leenhardt L, Clero D, Julien N, Venissac N, Tronc F, Dutau H, Marquette CH, Juvin C, Lebreton G, Cohen Y, Zogheib E, Beloucif S, Planes C, Tresallet C, Bensidhoum M, Petite H, Rouard H, Miyara M, Vicaut E. Airway replacement using stented aortic matrices: Long-term follow-up and results of the TRITON-01 study in 35 adult patients. Am J Transplant. 2022 Dec;22(12):2961-2970. doi: 10.1111/ajt.17137. Epub 2022 Jul 14. PMID 35778956